CLINICAL TRIAL: NCT03053856
Title: Phase II, Single-arm Study of Adjuvant Pembrolizumab in N2 Positive Non-small Cell Lung Cancer Treated With Neoadjuvant Concurrent Chemoradiotherapy Followed by Curative Resection
Brief Title: Adjuvant Pembrolizumab in N2 Positive Non-small Cell Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-09-018
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Stage IIIA Non-small Cell Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; Adjuvant pembrolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Cisplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: N2 positive stage IIIA non-small cell lung cancer treated with neoadjuvant concurrent chemoradiotherapy followed by curative resection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab arm (Experimental): Adjuvant Pembrolizumab
  Interventions: Drug: Pembrolizumab; Procedure: Curative resection; Procedure: Neoadjuvant concurrent chemoradiotherapy; Drug: Cisplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Adjuvant pembrolizumab 200 mg every 3 weeks for up to 24 months. (treated with neoadjuvant concurrent chemoradiotherapy followed by curative resection)
  Other Names: MK-3475
Procedure: Curative resection — Neoadjuvant concurrent chemoradiotherapy followed by curative resection
Procedure: Neoadjuvant concurrent chemoradiotherapy — RT 44 Gy/22 Fractions for 5 weeks With Chemotherapy (Cisplatin 25mg/m2 once weekly, Paclitaxel 50mg/m2 once weekly)
Drug: Cisplatin — 25mg/m2 once weekly
Drug: Paclitaxel — 50mg/m2 once weekly

SUMMARY:
This is a single arm, single center phase II study of adjuvant pembrolizumab in N2 positive non-small cell lung cancer (NSCLC) patients treated with neoadjuvant concurrent chemoradiotherapy followed by curative resection. Patients will receive pembrolizumab 200 mg every 3 weeks for up to 24 months.

The primary objective of this study is to assess the efficacy of adjuvant pembrolizumab treatment in terms of disease-free survival (DFS; per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 as assessed by the investigator).

The baseline assessment is part of the screening procedures and should be performed within 0 to 14 days before the start of study drug. The imaging modalities used for RECIST 1.1 assessment will be CT of chest or PET-CT if indicated. Follow-up chest CT for all patients will be assessed every 12 weeks for the first year, every 16 weeks for the second year, every 6 months for the third year, and every year thereafter. In subjects who discontinued study therapy without documented recurrence, every effort should be made to continue monitoring their disease status.

If an unscheduled assessment is performed, and the patient has not progressed, every attempt should be made to perform the subsequent assessments at their scheduled visits. RECIST 1.1 scans will be analyzed by the investigator on site; a central review will not be conducted.

Following completion or discontinuation of study drug, patients will enter a follow-up period.

Once a patient has had objective relapse recorded and has discontinued study drug, the patient will be followed for survival status every 3 months until death, withdrawal of consent or the end of the study.

Patients will also be requested to provide tumor samples from diagnostic (obtained before neoadjuvant CCRT) and surgical specimens for exploratory biomarker study. Sample provision is not optional, subject to a specific consent.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible for participation in this trial, the subject must:

  1. Be willing and able to provide written informed consent for the trial
  2. Be 18 years of age
  3. Be within 6 weeks after complete resection after neoadjuvant CCRT
  4. Have a performance status of 0 or 1 on the ECOG Performance Scale.
  5. Patients who completed neoadjuvant CCRT regimen includes 5 cycles of weekly Paclitaxel (50 mg/m2 + 5DW200 MIV over 1hr) plus Cisplatin (25 mg/m2 + N/S 150 mL MIV over 1hr) concurrent with radiotherapy (44 Gy/22fx daily fraction).
  6. Be willing to provide tissue from a obtained before neoadjuvant CCRT and surgical specimen (at least 10 slides from each surgically resected primary tumors and surgically resected metastatic lymph nodes)
  7. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days of treatment initiation.
  8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
  9. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

     Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
  10. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* The subject must be excluded from participating in the trial if the subject:

  1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
  2. Participation in another clinical study with PD-1 or PD-L1 inhibitors at any time
  3. Any previous treatment with a PD-1, PD-L1 inhibitor or any anti-cancer therapy after complete resection of lung cancer
  4. Current or prior use of immunosuppressive medication within 28 days before the first dose of pembrolizumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
  5. Mean QT interval corrected for heart rate (QTc) ≥470 ms using Bazett's correction
  6. Has a known history of active TB (Bacillus Tuberculosis)
  7. Active or prior documented inflammatory bowel disease (Crohn's disease or ulcerative colitis)
  8. History of allogenic organ transplant
  9. Hypersensitivity to pembrolizumab or any of its excipients.
  10. Prior history of malignancy within 2 years from study entry except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, or early gastric cancer. The incidentally detected, non-metastatic well differentiated thyroid cancer can be enrolled irrespective of the treatment, because the prognosis of this type of cancer is known much better than the study disease, even it is untreated. For the debatable double primary cancer, the enrolment can be discussed with the principal investigator in a manner of case by case, and if it is not expected to affect the study outcome, the subjects can be enrolled.
  11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  12. Has known history of, or any evidence of active, non-infectious pneumonitis.
  13. Evidence of interstitial lung disease.
  14. Has an active infection requiring systemic therapy.
  15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
  16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
  17. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
  18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
  19. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
  20. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2017-02-14 (Estimated); Primary Completion 2021-05-13 (Estimated); Study Completion 2021-08-13 (Estimated)

PRIMARY OUTCOMES:
Efficacy of adjuvant pembrolizumab in N2 Positive NSCLC | 24 months
  Disease free survival to evaluate the efficacy of adjuvant pembrolizumab in N2 positive non-small cell lung cancer patients treated with neoadjuvant concurrent chemoradiotherapy followed by curative resection.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of radomization until the date of death from any cause, withdrawal of consent, or the end of the study, assessed up to 120 months
  Pembrolizumab prolongs OS per RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015;372:2018-2028. — http://www.nejm.org/doi/full/10.1056/NEJMoa1501824
- See also: Global cancer statistics. CA Cancer J Clin. 2011;61:69-90. — https://www.ncbi.nlm.nih.gov/pubmed/21296855
- See also: The IASLC Lung Cancer Staging Project: proposals for the revision of the TNM stage groupings in the forthcoming (seventh) edition of the TNM Classification of malignant tumours. J Thorac Oncol. 2007;2:706-714. — https://www.ncbi.nlm.nih.gov/pubmed/17762336
- See also: Randomized trial of neoadjuvant therapy for lung cancer: interim analysis. Ann Thorac Surg. 1992;53:992-998. — https://www.ncbi.nlm.nih.gov/pubmed/1317697
- See also: A randomized trial comparing preoperative chemotherapy plus surgery with surgery alone in patients with non-small-cell lung cancer. N Engl J Med. 1994;330:153-158. — http://www.nejm.org/doi/full/10.1056/NEJM199401203300301
- See also: Mediastinal lymph node clearance after docetaxel-cisplatin neoadjuvant chemotherapy is prognostic of survival in patients with stage IIIA pN2 non-small-cell lung cancer: a multicenter phase II trial. J Clin O — https://www.ncbi.nlm.nih.gov/pubmed/12721251
- See also: Prognostic factors affecting long-term outcomes in patients with resected stage IIIA pN2 non-small-cell lung cancer: 5-year follow-up of a phase II study. Br J Cancer. 2006;94:1099-1106. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2361244/
- See also: Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012;366:2455-2465. — http://www.nejm.org/doi/full/10.1056/NEJMoa1200694
- See also: Acquired resistance to fractionated radiotherapy can be overcome by concurrent PD-L1 blockade. Cancer Res. 2014;74:5458-5468. — https://www.ncbi.nlm.nih.gov/pubmed/25274032